CLINICAL TRIAL: NCT03178526
Title: The Effect of Lovastatin Gel in the Treatment of Chronic Periodontitis Randomized Controlled Trial Split-mouth
Brief Title: The Effect of Lovastatin Gel in the Treatment of Chronic Periodontitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Islamic Azad University, Sanandaj (Other)
Responsible Party: Principal Investigator, Amirhossein Farahmand, The effect of lovastatin gel in the treatment of chronic periodontitis a randomized controlled trial with split-mouth, Islamic Azad University, Sanandaj
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 25187
Record Dates: First submitted 2017-06-05; First posted 2017-06-07 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Alveolar Bone Loss, Chronic Periodontitis, Lovestatin Gel, Regeneration
MeSH Terms: conditions — Alveolar Bone Loss; Chronic Periodontitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- levostatin gel (Active Comparator): levostatin gel 1.2% topical gel was put into teh periodontal pocket using an insulin syringe
  Interventions: Drug: Lovastatin gel
- placebo gel (Placebo Comparator): placebo gel 1.2% topical gel was put into the periodontal pocket using an insulin syringe
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lovastatin gel — Lovastatin gel1.2% topical gel was put into teh periodontal pocket using an insulin syringe
  Other Names: Group A
  Arms: levostatin gel
Drug: Placebo — placebo gel
  Arms: placebo gel

SUMMARY:
Aim: dis double-blind split-mouth clinical trial study was performed to evaluate teh clinical and radiographic effect of local delivery of lovastatin gel as an adjunct to scaling and root planning (SRP) in teh treatment of chronic periodontitis.

Method and Materials: 15 patients with two mandibular molar teeth with probing depth (PD)≥3 mm, clinical attachment level (CAL)≥3 mm and bone loss more than 3 mm according to parallel periapical x-ray and distance from CEJ to alveolar crest, were selected.Totally 24 mandibular molars were selected for teh study.

Clinical periodontal parameters included PD, CAL, bleeding index(BI), plaque index(PI) were recorded for teh selected teeth at baseline and at 1,3 and 6 months. Radiographic assessments were performed at baseline and after 6 months. At one side teh pockets around randomly selected molar were injected with a blunt syringe filled with lovastatin gel 1.2%( case group=B), and on teh other side, teh pockets were filled with a placebo gel by a blunt syringe ( control group=A).Two-way repeated measure ANOVA test and T-test were used for statistic analysis Spss 23.( P<0.05) was considered significant.

DETAILED DESCRIPTION:
Statins are an important group of hypolipidemic drugs dat are able to modulate inflammation and alveolar bone loss. Rosuvastatin (RSV) and atorvastatin (ATV) are non to inhibit osteoclastic bone resorption and has been proposed to has osteostimulative properties.

ELIGIBILITY:
Inclusion Criteria:

24 patients wif periodontitis chronic and TEMPhas a 2 molar symmetrically in the lower jaw pockets of periodontal depth of at least 4 mm and CAL greater than 3 mm in at least one of the surfaces of the teeth, the X-ray bars from both sides of the molar regions jaw bottom, from CEJ and alveolar crest was more than 3 mm, were selected

Exclusion Criteria:

1. systemic disease
2. pregnancy or breastfeeding
3. allergy drug used
4. smoking
5. medication 6. not willing to consent to participate in the study

7-Trismus 8-The type of disease periodontal (Aggressive) 9. History of periodontal treatment in the previous 6 months 10-orthodontic treatment

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2015-12-24 (Actual); Primary Completion 2016-01-13 (Actual); Study Completion 2016-02-13 (Actual)

PRIMARY OUTCOMES:
Bone defect fill | Three months
  radiographic analysis for bone defect

IPD SHARING:
Plan to Share IPD: No